CLINICAL TRIAL: NCT06489028
Title: A Pivotal, Randomized, Placebo-controlled, Double-blind, Multicenter, International Phase III Clinical Trial to Investigate the Efficacy and Safety of Allo-APZ2-CVU on Wound Healing of Therapy-Resistant Non-Healing Chronic Venous Ulcers (CVU)
Brief Title: Allogeneic ABCB5-positive Dermal Mesenchymal Stromal Cells for Treatment of Therapy-resistant CVU (Phase III)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: RHEACELL GmbH & Co. KG (Industry)
Collaborators: FGK Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: allo-APZ2-CVU-III; 2024-512720-11-00 (EU CTIS Number); U1111-1305-5114 (Registry Identifier: World Health Organization [WHO] Registry Network)
Record Dates: First submitted 2024-06-25; First posted 2024-07-05 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Venous Leg Ulcer
Keywords: Chronic Venous Ulcer; ABCB5; Allogeneic; Dermal mesenchymal stromal cells; varicose ulcer; skin ulcer; advanced therapy medicinal product; somatic cell therapy; phase III
MeSH Terms: conditions — Varicose Ulcer; Skin Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Verum (Experimental)
  Interventions: Drug: allo-APZ2-CVU
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: allo-APZ2-CVU — Allogeneic dermal ABCB5-positive Mesenchymal Stromal Cells (ABCB5+ MSCs)
  Arms: Verum
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The aim of this clinical trial is to investigate the efficacy and safety of allo-APZ2-CVU, administered topically on therapy-resistant non-healing CVUs compared to placebo.

DETAILED DESCRIPTION:
This is a pivotal, randomized, placebo-controlled, double-blind, multicenter, international phase III clinical trial to investigate the efficacy and safety of the IMP allo-APZ2-CVU on wound healing in patients with therapy-resistant non-healing CVU.

The allogeneic IMP allo-APZ2-CVU contains skin-derived ABCB5-positive dermal mesenchymal stromal cells isolated from skin tissue of healthy donors and stored in a donor cell bank.

Patients will be randomized to be treated with allo-APZ2-CVU or placebo. The patients will undergo treatment with the IMP on Day 0 (V3) and will be followed up for efficacy for 18 weeks (V4 until V14). Three safety follow-up visits will be performed at Month 6 (V15), Month 10 (V16) and Month 16 (V17).

The wound healing process will be documented by standardized photography.

The wound size measurement will start at the first Screening Visit (V1) and will be measured at each following on-site visit.

Pain will be assessed using a numerical rating scale and quality of life will be investigated with standardized and validated questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Patients at least 18 years old;
2. Chronic venous leg ulcer at lower leg and/or ankle region that has not been present longer than 15 years, diagnosed by Doppler or Duplex sonography, ankle brachial index, physical examination and dermatological review;
3. Wound size at V1 and V2 between 1 and 25 cm˄2 as measured by standardized photography;
4. If patients have 2 or more ulcers at the same extremity, the target ulcer has to be separated from the other ulcers with a bridge of epithelialized skin at least 1 cm wide;
5. Body mass index between 15 and 50 kg/m²;
6. Patients able to understand the nature of the study and able to provide written informed consent prior to any clinical trial procedures;
7. Women of childbearing potential must have a negative urine pregnancy test at Visit 1;
8. During the course of the clinical trial women of childbearing potential and their male partners must be willing to use highly effective contraceptive methods as defined in the EMA CTCG "Recommendations related to contraception and pregnancy testing in clinical trials" Version 1.2.

Exclusion Criteria:

1. Evidence of the ulcer extending to the underlying muscle, tendon, or bone;
2. Uncontrolled Diabetes mellitus i.e. Hemoglobin A1c (HbA1c) >9.0% (75 mmol/mol) (measured by blood test);
3. Peripheral Artery Disease including claudication with need of treatment or intervention;
4. Acute deep vein thrombosis diagnosed within 30 days before V1, or untreated deep vein thrombosis;
5. Wounds showing size reduction of more than 40% at Visit 2 compared to Visit 1;
6. Patients with known hypersensitivity and/or clinical contraindications to the compression systems used in the clinical trial, or inability/unwillingness to tolerate leg ulcer compression systems;
7. Acute wound infection of ulcer requiring treatment as judged clinically;
8. Current use of medications that are known to influence wound healing i.e. systemic immunosuppressives, cytotoxic medicinal products, systemic steroids (above Cushingthreshold level) at investigator´s discretion;
9. Patients who, in the opinion of the investigator, for any reason are unable or unwilling to complete the trial per protocol (e.g. alcohol or substance abuse, not mobile, short life expectancy) or there is an evidence of any other medical condition (such as psychiatric illness, physical examination, or laboratory findings) that may interfere with the planned treatment, affect the patient's compliance, or place the patient at high risk of complications related to the treatment;
10. Any malignancy within the past 5 years, excluding successfully treated carcinoma in situ, basal cell carcinoma or squamous cell carcinoma of the skin without evidence of metastases;
11. Pregnant or lactating women;
12. Known hypersensitivities to the active substance or to any of the excipients in the IP or the placebo;
13. Surgical procedure affecting the CVU, such as bypass or mesh graft performed within two months prior to Visit 1;
14. Current or previous (within 30 days of enrollment) treatment with another IP, or participation in another clinical trial, including follow-up phase;
15. Previous participation in this clinical trial (except for screening failures due to an inclusion or exclusion criterion);
16. Employees of the sponsor, or employees or relatives of the investigator(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-12-26 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Complete wound closure | 18 weeks
  Complete wound closure already persisting for at least two weeks

SECONDARY OUTCOMES:
Complete wound closures at each post-baseline follow-up visit | at each post-baseline follow-up visit (starting the day after intervention until month 16)
  Complete wound closures at each post-baseline follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Anna Moessmer, Study Director — RHEACELL GmbH & Co. KG
Locations (15):
- United States (4):
  - RHEACELL Clinical Trial Site, Hialeah, Florida
  - RHEACELL Clinical Trial Site, Miami, Florida
  - RHEACELL Clinical Trial Site, Boston, Massachusetts
  - RHEACELL Clinical Trial Site, Minneapolis, Minnesota
- RHEACELL Clinical Trial Site, Multiple Locations, Austria
- RHEACELL Clinical Trial Site, Multiple Locations, Czechia
- RHEACELL Clinical Trial Site, Multiple Locations, France
- RHEACELL Clinical Trial Site, Several Locations, Germany
- RHEACELL Clinical Trial Site, Multiple Locations, Hungary
- RHEACELL Clinical Trial Site, Multiple Locations, Italy
- RHEACELL Clinical Trial Site, Multiple Locations, Netherlands
- RHEACELL Clinical Trial Site, Multiple Locations, Poland
- RHEACELL Clinical Trial Site, Multiple Locations, Slovakia
- RHEACELL Clinical Trial Site, Multiple Locations, Sweden
- RHEACELL Clinical Trial Site, Multiple Locations, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided